CLINICAL TRIAL: NCT06604520
Title: Functional Neuroimaging to Examine Affective Symptoms and Cognition in Frontotemporal Dementia
Brief Title: Vortioxetine for the Treatment of Mood and Cognitive Symptoms in Frontotemporal Dementia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Lundbeck LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00403796; 1K23AG088248 (NIH)
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Fronto-temporal Dementia; Fronto-temporal Lobar Dementia; Frontotemporal Degeneration; Frontotemporal Dementia (FTD); Frontotemporal Dementia, Behavioral Variant; Frontotemporal Dementia
Keywords: FTD; Frontotemporal Dementia; Neuropsychiatric Symptoms; Antidepressant
MeSH Terms: conditions — Frontotemporal Dementia; Pick Disease of the Brain | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patient Treatment Arm (Vortioxetine) (Experimental): Individuals with bvFTD and mood symptoms receiving the study drug, vortioxetine.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Individuals with bvFTD and mood symptoms will receive approximately 12 weeks of treatment with vortioxetine
  Other Names: Trintellix

SUMMARY:
The goal of this clinical trial is to learn if vortioxetine improves mood symptoms and cognition in patients with early-stage behavioral variant Frontotemporal Dementia (bvFTD). The main questions this study aims to answer are:

1. Do individuals with mood symptoms and bvFTD have brain changes and cognitive profiles that differ compared to individuals without bvFTD?
2. Do mood symptoms and cognition improve following treatment with vortioxetine?

Researchers will also determine whether there are changes in the brain associated with vortioxetine treatment.

Participants will:

* Undergo a screening visit that involves clinical assessments and laboratory tests
* Undergo an initial brain magnetic resonance imaging (MRI) and fluorodeoxyglucose (18F) Positron Emission Tomography (FDG PET) scan before starting treatment with vortioxetine
* Undergo memory and problem-solving tests before starting treatment with vortioxetine
* Undergo approximately 12 weeks of treatment with vortioxetine, during which time there will be regular contact and assessments with the study psychiatrist
* Undergo a repeat PET scan and repeat memory and problem-solving tests after 12 weeks of treatment with vortioxetine

ELIGIBILITY:
FTD Patients

Inclusion Criteria:

1. Male or Female
2. Age 45 and above
3. Diagnosis of possible or probable bvFTD based on international consensus criteria for behavioral variant FTD (FTDC)
4. The presence of at least one of the following affective symptoms on the 12-item Neuropsychiatric Inventory: depression, anxiety, irritability, or agitation
5. A global Clinical Dementia Rating (CDR®) plus National Alzheimer's Coordinating Center (NACC) Frontotemporal lobar degeneration (FTLD) Behavior and Language Domains global score (CDR® plus NACC FTLD) less than or equal to one
6. Patients must be medically stable
7. Vortioxetine treatment is clinically indicated
8. Competent to provide informed consent

Exclusion Criteria:

1. No history of drug or alcohol dependence within six months prior to study entry
2. Negative toxicology screening for drugs of abuse
3. Subject must not be pregnant or nursing
4. No contraindications to Vortioxetine treatment
5. No contraindications for Magnetic Resonance (MR) scanning (e.g. metal implanted in the body)

Healthy Controls

Inclusion Criteria:

1. Male or Female
2. Age 45 and above
3. Subjects must be medically stable
4. Free of psychotropic medications
5. Competent to provide informed consent

Exclusion Criteria:

1. No current or past history of neurological or psychiatric illness or substance abuse
2. Subject must not be pregnant or nursing
3. Negative toxicology screening for drugs of abuse
4. No contraindications for MR scanning (e.g. metal implanted in the body)

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in global cerebral glucose metabolism on [18F] fluorodeoxyglucose Positron Emission Tomography (FDG PET) | Baseline, 12 weeks
  Cerebral glucose uptake measured through 18F FDG positron emission tomography

SECONDARY OUTCOMES:
Change in depressive symptoms as assessed by the Hamilton Depression Rating Scale (HDRS). | Baseline, 12 weeks
  The HDRS is a widely used clinician-administered depression assessment tool designed to measure the severity of depression in individuals. It consists of 17 items rated on a 3 or 5 point scale with total scores ranging from 0 to 52. A higher score indicates more severe symptoms of depression.

OTHER OUTCOMES:
Change in performance on the Trail Making Test (TST). | Baseline, 12 weeks
  The TMT is a widely used neuropsychological test that assesses an individuals cognitive abilities including executive function, attention, processing speed, and mental flexibility. It is divided into two parts: Trail Making Test A and Trail Making Test B. The Trail Making Test A primarily assesses visual attention and processing speed. Time taken to complete the task is recorded, with faster times indicating better cognitive performance. The Trail Making Test B primarily assesses cognitive flexibility, executive functioning, task switching and attention. Time taken to complete the task is recorded, with faster times indicating better cognitive performance.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Morrow, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data will be preserved and shared in the National Archive of Computerized Data on Aging (NACDA).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will shared 12 months after study starts and every 6 months thereafter. All data will be shared upon publication or at the end of the award period, whichever is sooner. For published studies, data will be shared when the pre- print is available. NACDA studies have digital object identifiers (DOI) to aid in findability. The investigators will include that DOI in relevant publications. NACDA will make decisions about how long to preserve the data, but that data archive has not deleted any deposited data up to now.
Access Criteria: Given that all data will be de-identified, the investigators do not plan to control access to the data or require a Data Use Agreement. Data submitted to NACDA that are evaluated as constituting a low disclosure risk are publicly released and available to download directly from the NACDA website. The investigators plan to prepare and submit the data in a de-identified format in order to minimize any disclosure risk and allow for public release through NACDA. NACDA performs an evaluation of all submitted data prior to release to ensure disclosure risks are minimized, and the investigators anticipate approval for public release of data without restriction through the NACDA website.
URL: https://www.icpsr.umich.edu/web/pages/NACDA/index.html